CLINICAL TRIAL: NCT03076060
Title: Randomised Controlled Crossover Double-blind Study on Very Low Calories Ketogenic Diet in Overweighted Migraine Patients.
Brief Title: Very Low Calories Ketogenic Diet in Migraine.
Acronym: Ketomig
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Cherubino DI LORENZO, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChEmicrania
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Migraine; Overweight and Obesity
Keywords: Ketogenic Diet; Very low calories diet; ketone bodies
MeSH Terms: conditions — Migraine Disorders; Overweight; Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraineurs (Experimental): Overweighted or Obese migraineurs that refer to a dietician clinic to treat their ponderal condition.
  Intervention: 4-week of VLCKD by meal replacements poor in fats and carbohydrates.
  Interventions: Behavioral: Ketogenic diet
- Sham diet migraineurs (Sham Comparator): Overweighted or Obese migraineurs that refer to a dietician clinic to treat their ponderal condition.
  Intervention: 4-week of non-ketogenic VLCD by meal replacements poor in fats and proteins.
  Interventions: Behavioral: Sham Diet

INTERVENTIONS:
Behavioral: Ketogenic diet — Two different kind of diet, a Very Low Calories Ketogenic Diet (KD) and a sham weight-loss diet (SD), will be consecutively administered in each patient recruited in the study for one month. To avoid the bias of different caloric intake, SD group will undergo to a non-ketogenic Very Low Calories Diet . Randomly patients will start with KD or SD.
  Patients assigned to this arm will follow the KD.
  Other Names: Very Low Calories Ketogenic Diet
  Arms: Migraineurs
Behavioral: Sham Diet — Two different kind of diet, a Very Low Calories Ketogenic Diet (KD) and a sham weight-loss diet (SD), will be consecutively administered in each patient recruited in the study for one month. To avoid the bias of different caloric intake, SD group will undergo to a non-ketogenic Very Low Calories Diet . Randomly patients will start with KD or SD.
  Patients assigned to this arm will follow the SD.
  Other Names: Non-Ketogenic Very Low Calories Diet
  Arms: Sham diet migraineurs

SUMMARY:
Ketogenesis is a physiologic phenomenon due to starvation or ketogenic diet (KD), a drastic restricted carbohydrate dietary regimen that induces lipid metabolism and ketone body (KB) synthesis. We followed, in a dietician clinical setting, a group of migraineurs who randomly received a one-month prescription of experimental diet, followed by a one-month of carbohydrate progressive reintroduction, then another one-month of experimental diet, followed by a one-month of carbohydrate progressive reintroduction. Experimental diets are a very-low calorie KD, or an isocaloric non-ketogenic diet.

Aim of our study is verify if during ketogenesis migraine improves.

DETAILED DESCRIPTION:
The ketogenic diet (KD) is a high-fat, low-carbohydrate diet for long used to treat refractory epilepsy. Ketogenesis, ketone-body formation, is a physiologic phenomenon also observed in patients following low-carbohydrate low-calorie diets for rapid weight loss. Different Authors evidenced a protective effect of ketone bodies also on migraine; however, KD effectiveness in this disorder is under scrutiny yet again. In fact, some concerns makes the matter a still open question: available studies were anecdotal, or conducted on small numbers; not all patients were diagnosed as migraineurs according to current headache classification; during ketogenesis there could be an avoidance of potentially trigger foods. Moreover, to comply with ketogenic diet, great motivation is needed and often migraineurs did not have it.

Aim of this study is verify in a double blind parallel group cross over design if ketogenesis is really able to prevent/avoid headache attacks in episodic migraineurs.

Methods: Thirty-five consecutive episodic migraineurs, with an attack frequency higher than 2 attacks per months, will be enrolled. Two different kind of diet, a KD and a standard weight-loss diet (SD), will be consecutively administered in each patient recruited in the study for one month. Randomly patients will start with KD or SD. At the end of the second month differences between diets will be detected.

KD will consist of 4 daily pharmaceutical meal substitutes composed by low-carbohydrate, low-fat, rich in protein serving of food, already commercially available. SD will consist in a similar eating program, with serving of food with addition of carbohydrate to avoid ketogenesis.

ELIGIBILITY:
Inclusion Criteria:

* kept a headache diary for at least 1 month
* migraine disease onset before the age of 50
* at least one migraine attack per month in the last 3 months
* <15 days/month with headaches.

Exclusion Criteria:

* prophylactic treatment in the previous 3 months
* over consumption of acute anti-migraine medication (triptan, analgesic, or ergotamine)
* pregnancy or lactation
* type I diabetes
* serious organic or psychiatric disorders that the investigators judged as having the potential to influence the trial evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Migraine attacks frequency | one-month
  number of attacks per month

SECONDARY OUTCOMES:
Migraine days | one-month
  number of days with migraine per month
Drug consumption | one-month
  number of symptomatic drugs assumed per month to treat migraine

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pierelli, Study Director — Sapienza Univeristy
Locations (1):
- Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
We do not share data.

REFERENCES:
- [Result] Di Lorenzo C, Coppola G, Sirianni G, Di Lorenzo G, Bracaglia M, Di Lenola D, Siracusano A, Rossi P, Pierelli F. Migraine improvement during short lasting ketogenesis: a proof-of-concept study. Eur J Neurol. 2015 Jan;22(1):170-7. doi: 10.1111/ene.12550. Epub 2014 Aug 25. PMID 25156013